CLINICAL TRIAL: NCT00702884
Title: A Mechanistic Radiographic and Biologic Phase 2 Single Agent Study of Sunitinib Malate in Relapsed/Refractory Esophageal and Gastroesophageal Cancers
Brief Title: Sunitinib in Treating Patients With Relapsed or Refractory Esophageal or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tony Bekaii-Saab (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07121; NCI-2011-03148 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Esophageal Cancer
Keywords: recurrent esophageal cancer; stage IIIA esophageal cancer; stage IIIB esophageal cancer; stage IIIC esophageal cancer; stage IV esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Sunitinib 37.5 mg daily for a 4 week cycle
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Sunitinib 37.5 mg daily for a 4 week cycle
  Other Names: Sutent; SU011248 L-Malate salt; SU010398; PHA-290940AD; SU011248

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with relapsed or refractory esophageal or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the progression-free survival rate (complete response, partial response, and stable disease as defined by RECIST criteria [Response Evaluation Criteria in solid Tumors]) at 24 weeks in patients with relapsed or refractory esophageal or gastroesophageal junction cancer treated with sunitinib malate.

Secondary

* To explore the predictive role of a hybrid imaging protocol that combines PET/CT (Positron emission tomography) scan simultaneously with dynamic contrast-enhanced MRI.
* Correlate quantitative changes in mean vessel density, alterations in tumor cell proliferation, and apoptosis in tumor biopsy specimens with clinical outcome in these patients.
* To evaluate the objective response as defined by RECIST criteria, median overall survival, and median progression-free survival of these patients.
* To evaluate the toxicities of sunitinib malate in these patients.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and tumor tissue sample collection periodically for correlative laboratory studies. Tumor tissue samples are assessed by immunohistochemistry and TUNEL for detection and quantitation of mean vessel density, proliferating tumor cells, and apoptosis. Tumor tissue samples are also assessed by immunohistochemistry for MAPK levels. Blood samples are analyzed by ELISA for VEGF, PlGF, sVEGFR2, and sVEGFR3 levels. Patients also undergo PET/CT scan and dynamic contrast-enhanced MRI periodically for correlative studies.

After completion of study treatment, patients are followed for at least 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed esophageal or gastroesophageal junction carcinoma that is not amenable to curative surgery or other curative therapy

  * Advanced, relapsed or refractory disease
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* No known brain metastases

PATIENT CHARACTERISTICS:

* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Life expectancy > 12 weeks
* WBC ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Serum calcium ≤ 12.0 mg/dL
* Total bilirubin normal
* AST (aspartate aminotransferase) and ALT (Alanine Aminotransferase) ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for 28 days after completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* No ongoing cardiac dysrhythmias ≥ grade 2, atrial fibrillation of any grade, or prolongation of the QTc (corrected QT interval) interval to > 450 msec (for males) or > 470 msec (for females)
* No hypertension that cannot be controlled by medications (i.e., systolic/diastolic blood pressure > 150/100 mm Hg despite optimal medical therapy)
* No myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 12 months
* No cerebrovascular accident or transient ischemic attack within the past 12 months
* No pulmonary embolism within the past 12 months
* No condition that would impair the ability to swallow and retain sunitinib malate tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease)
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No serious or nonhealing wound, ulcer, or bone fracture
* No pre-existing thyroid abnormality that cannot be maintained in the normal range with medication
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* At least 4 weeks since prior radiotherapy or major surgery
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin C, carmustine, or alkylating agents)
* No more than 6 prior courses of an alkylating agent
* No more than 450 mg/m² of prior doxorubicin hydrochloride or 900 mg/m² of prior epirubicin hydrochloride
* No more than 2 lines of prior therapy in the metastatic setting
* No prior anti-VEGF monoclonal antibodies, such as bevacizumab or aflibercept
* No prior tyrosine kinase inhibitors with similar targets (e.g., sorafenib tosylate or axitinib)
* No other concurrent investigational agents
* No concurrent therapeutic doses of coumarin-derivative anticoagulants, such as warfarin

  * Warfarin at doses of ≤ 2 mg daily are allowed for prophylaxis of thrombosis
  * Low molecular weight heparin allowed provided PT/INR (Prothrombin time and international normalized ratio) is ≤ 1.5
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent agents with proarrhythmic potential (e.g., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2013-09-17 (Actual); Study Completion 2013-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Wu C, Mikhail S, Wei L, Timmers C, Tahiri S, Neal A, Walker J, El-Dika S, Blazer M, Rock J, Clark DJ, Yang X, Chen JL, Liu J, Knopp MV, Bekaii-Saab T. A phase II and pharmacodynamic study of sunitinib in relapsed/refractory oesophageal and gastro-oesophageal cancers. Br J Cancer. 2015 Jul 14;113(2):220-5. doi: 10.1038/bjc.2015.197. Epub 2015 Jul 7. PMID 26151457
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sunitinib
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years] | 61 [38 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 22
Race/Ethnicity, Customized [Number; unit: patients]
  White | 23
  Black | 2
Region of Enrollment [Number; unit: patients]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate
Description: Complete response, partial response, and stable disease) as assessed by RECIST criteria at 24 weeks
Time Frame: up to 24 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
weeks | 7 [5.6 to 11.4]

2. Secondary Outcome: Overall Response Rate
Description: The Overall Response Rate (ORR) was assessed using Partial Response + Complete Response for patients. Response and progression was evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0.
Time Frame: up to 4 years
Population: Durable Complete Response= PR + SD > 10 weeks
Measure: Number; unit: patients
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
patients | 10

3. Secondary Outcome: Median Overall Survival Time
Description: The median overall survival time will be reported using the 95% confidence intervals for the parameters.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
weeks | 16.6 [8.9 to 25.3]

4. Secondary Outcome: Median Progression-free Survival Time
Description: Progression free survival was measured as the time from start of treatment to the first measurement of tumor growth.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 25
weeks | 6.9 [5.6 to 11.4]

5. Secondary Outcome: Frequency and Severity of Adverse Events
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was utilized for adverse event reporting.
Time Frame: up to 4 years
Measure: Number; unit: percentage of patients
Groups:
- Grade 1 and 2 Adverse Events: Grade 1=Mild; asymptomatic or mild symptoms
  Grade 2=Moderate; minimal, local or noninvasive intervention indicated
- Grade 3 Adverse Events: Grade 3=Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated
- Grade 4 Adverse Events: Grade 4=Life-threatening consequences; urgent intervention indicated
Arm/Group | Grade 1 and 2 Adverse Events | Grade 3 Adverse Events | Grade 4 Adverse Events
Number analyzed (Participants) | 25 | 25 | 25
percentage of patients
  Fatigue | 52 | 24 | 0
  Anemia | 48 | 12 | 8
  Thrombocytopenia | 12 | 12 | 4
  Leukopenia | 32 | 12 | 4

6. Secondary Outcome: Change in Mean Vessel Density
Description: Quantitative assessment of proliferating tumor cells, and apoptosis, of the laboratory and radiographic correlates, the analyses will be purely explorative.
Time Frame: up to 4 years
Population: Insufficient tissue was available and the analysis for mean vessel density not performed
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

7. Secondary Outcome: Quantitative Assessment of Proliferating Tumor Cells and Apoptosis
Description: Biopsy sample taken from patients before and after treatment Apoptosis measures using the terminal deoxynucleotidyl transferase-mediated dUTP nick end labeling (TUNEL) assay, which measures 3' nicked DNA. DNA is degraded in the early steps of apoptosis into low molecular weight (LMW) fragments and the production of single strand breaks in the high molecular weight DNA.Both of these features of apoptosis can be detected by labeling free 3'-OH termini with modified nucleotides, in our case this will be biotin-labeled dUTP. Terminal deoxynucleotidyl transferase (TdT) is an enzyme that labels blunt-ends of DNA breaks and can catalyze polymerization of nucleotides to free 3'-OH DNA ends in a template-independent manner. The newly incorporated nucleotides are detected by a secondary antibody, avidin-peroxidase. After substrate reaction, the stained cells can be detected and counted under a light microscope. Apoptotic cells will be fixed with formaldehyde which links LMW DNA
Time Frame: up to 4 years
Population: Analysis for tumor cells not performed due to insufficient samples available
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Toxicities were graded according to NCI Common Toxicity Criteria version 3.0
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 25/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=25)
Fatigue (General disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
GI Hemorrhage (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Hypertension (Vascular disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 8 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=25)
Leukopenia (Investigations) | 10 (10)
Lymphopenia (Investigations) | 7 (7)
Neutropenia (Investigations) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Thrombocytopenia (Injury, poisoning and procedural complications) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Fatigue (General disorders) | 15 (15)
Mucositis (Gastrointestinal disorders) | 7 (7)
Hypertension (Vascular disorders) | 2 (2)
GI Hemorrhage (Gastrointestinal disorders) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less